CLINICAL TRIAL: NCT01893632
Title: Gabapentin Treatment of Benzodiazepine Dependence
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient recruitment, funding terminated from sponsor
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, John Mariani MD, Assistant Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6740
Record Dates: First submitted 2013-06-29; First posted 2013-07-09 (Estimated); Results first posted 2018-07-24 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Benzodiazepine Dependence
Keywords: Benzodiazepines; clonazepam; alprazolam; Klonopin; Xanax; diazepam; Valium; lorazepam; Ativan
MeSH Terms: interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gabapentin (Experimental): All study medication will be over-capsulated with riboflavin to assess compliance using quantitative fluoroscopy. All participants will take three capsules three times per day throughout the study period. During week 1, GBP will be titrated over a five-day period to the dose target (GBP 1200 mg three times daily) or the maximum tolerated dose. Medication dosing will continue at GBP 1200 mg three times daily or placebo through the end of the study period (week 12). Dose reductions will be made for tolerability if necessary.
  Interventions: Drug: gabapentin
- Placebo (Placebo Comparator): Capsules filled with riboflavin.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: gabapentin
  Other Names: Neurontin
  Arms: Gabapentin
Drug: Placebo
  Arms: Placebo

SUMMARY:
Benzodiazepine dependence is a growing public health problem for which very few evidenced-based treatment approaches are available. Approximately 683,000 individuals met past year criteria for sedative-hypnotic use disorders in the US during 2010, a prevalence greater than heroin or methamphetamine dependence. The most commonly prescribed sedative-hypnotic agents are the benzodiazepines. Chronic use induces pharmacodynamic tolerance in the GABA neurotransmitter system and individuals with physiological dependence find benzodiazepines difficult to discontinue because of withdrawal or rebound symptoms, which include autonomic arousal, depression, anxiety, and insomnia. Available evidence-based treatment approaches have been primarily directed at therapeutic users of benzodiazepines who do not meet criteria for a substance use disorder, with a general consensus that the gradual taper of benzodiazepines over a period of several months is the optimal approach. However, patients with benzodiazepine dependence are typically referred for inpatient detoxification treatment, which rapidly tapers patients off benzodiazepines. Protracted withdrawal symptoms frequently persist after discharge, predisposing patients to relapse. More effective pharmacotherapeutic strategies are needed for the treatment of benzodiazepine dependence in the outpatient setting.

DETAILED DESCRIPTION:
Gabapentin has proven to be a safe and well-tolerated medication with a low abuse liability, thereby making it ideal for use in the outpatient setting.

The proposed Exploratory Development research project is a double-blind randomized controlled clinical trial comparing the efficacy of gabapentin to placebo for the outpatient treatment of benzodiazepine dependence. The goal of this project is to study the effects of gabapentin on the participants' benzodiazepine use in a facilitated taper-to-abstinence model, where participants will be actively using benzodiazepines at study entry, gabapentin treatment will be introduced, and participants will be counseled to gradually discontinue benzodiazepine use over the study period while gabapentin treatment is maintained. A modified version of Medical Management will be used to facilitate compliance with study medication and other study procedures, and includes clinical instruction for gradually reducing benzodiazepine use 25% per week. Benzodiazepines are not prescribed in the proposed study; participants continue to obtain benzodiazepines from their own prescribed or nonprescribed sources.

ELIGIBILITY:
Inclusion Criteria:

1. Meets DSM-IV-TR criteria for BZD dependence
2. Using BZDs a minimum of 5 days per week over the past 28 days
3. Between the ages of 18 and 60
4. Able to provide informed consent

Exclusion Criteria:

1. Any current DSM-IV-TR Axis I psychiatric disorder, other than BZD dependence, that might require intervention over the course of the study, including schizophrenia, bipolar disorder, major depressive disorder or panic disorder.
2. Receiving psychotropic medication other than BZDs
3. Evidence of physiological BZD withdrawal (pulse > 100; blood pressure > 140/90)
4. History of BZD withdrawal seizures or withdrawal delirium
5. History of allergic reaction to GBP
6. Pregnancy, lactation, or failure in female patients to use adequate contraceptive methods
7. Unstable physical disorders which might make participation hazardous medical history
8. Subjects who have a current DSM-IV-TR diagnosis of other substance dependence, with the exception of nicotine and caffeine history; dependence

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2016-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John J. Mariani, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- John Mariani, New York, New York, United States

REFERENCES:
- See also: Study Website — http://stars.columbia.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Gabapentin: All study medication will be over-capsulated with riboflavin to assess compliance using quantitative fluoroscopy. All participants will take three capsules three times per day throughout the study period. During week 1, GBP will be titrated over a five-day period to the dose target (GBP 1200 mg three times daily) or the maximum tolerated dose. Medication dosing will continue at GBP 1200 mg three times daily or placebo through the end of the study period (week 12). Dose reductions will be made for tolerability if necessary.
  gabapentin
- Placebo: Capsules filled with riboflavin.
  Placebo
Period: Overall Study
Arm/Group | Gabapentin | Placebo
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Placebo | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (0) | 59 (0) | 59 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Abstinence From Benzodiazepine Use
Description: Achievement of two weeks abstinence from benzodiazepine use at end of trial
Time Frame: last two weeks of 12 week trial
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks of trial
Arm/Group | Gabapentin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin (N=1) | Placebo (N=1)
anxiety (General disorders) | 0 (0) | 1 (1)
appetite change (Gastrointestinal disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
unsteady gait (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
chest tightness (General disorders) | 0 (0) | 1 (1)
confusion (General disorders) | 1 (1) | 0 (0)
coordination issues (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
sensory overstimulation (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
due to poor recruitment, enrollment was limited to two participants and trial was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes